CLINICAL TRIAL: NCT02594540
Title: Effects of the Mechanical Peripheral Stimulation for Parkinson's Disease Rehabilitation - A Randomized Clinical Trial
Brief Title: Effects of the Mechanical Peripheral Stimulation for Parkinson's Disease Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Gondola Medical Devices (Unknown); Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APA2016
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feet Mechanical Stimulation (Experimental): The feet mechanical stimulation will be given to all participants using GONDOLA equipment (Ecker Technologies Sagl, Switzerland). Intervention: Device: Foot Mechanical Stimulation (GONDOLA)
  Interventions: Device: Mechanical Peripheral Stimulation (GONDOLA)
- Sham Feet Mechanical Stimulation (Sham Comparator): The sham stimulation will be given to all participants using GONDOLA equipment (Ecker Technologies Sagl, Switzerland). Intervention: Device: Foot Mechanical Stimulation (GONDOLA)
  Interventions: Device: Mechanical Peripheral Stimulation (GONDOLA)

INTERVENTIONS:
Device: Mechanical Peripheral Stimulation (GONDOLA)
  Other Names: GONDOLA equipment (Ecker Technologies Sagl, Switzerland)

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of the peripheral mechanical stimulation of the feet on gait variables, clinical status, risk of falls, BDNF levels, immunological profile and brain functional connectivity changes in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Patients will be submitted to 8 sessions of peripheral mechanical stimulation of the feet or sham stimulation along 4 weeks.

Evaluations will be performed before and after the first session, after the forth and the eighth session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease based on clinical criteria, dopamine transporter (DaT) scans and/or magnetic resonance imaging;
* Able to walk 25 feet unassisted or with minimal assistance;
* Presenting freezing of gait;
* Aged between 50-85 years;
* Minimum score of 20 in the Mini Mental State Examination (MMSE);

Exclusion Criteria:

* Secondary musculoskeletal disorder involving the lower limb, as chondral injuries, ligament and ankle sprains which may impede the realization of the gait by pain or motion disability;
* Peripheral neuropathy;
* Not attending all the treatment;
* Absolute contraindications for fMRI (just for fMRI examination);
* Presence of deep brain stimulation;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Kinetic and kinematic gait analysis | 4 weeks of treatment
  Evaluated by means of the 3-D motion analysis system (BTS SMART DX 400).

SECONDARY OUTCOMES:
Risk of falls | 4 weeks of treatment
  Evaluated by means of the Timed Up & Go Test (TUG).
Motor impairment | 4 weeks of treatment
  Evaluated by means of the Unified Parkinson Disease Rating Scale (UPDRS III).
Level of depression | 4 weeks of treatment
  Evaluated by means of the Beck Depression Inventory (BDI).
Symptoms of Parkinson's disease progress | 4 weeks of treatment
  Evaluated by means of the Hoehn and Yahr scale.
Serum levels of BDNF | 4 weeks of treatment
  Analyzed in blood sampling.
Sensorio-motor connectivity | 4 weeks of treatment
  Functional magnetic resonance imaging.
Lymphocyte Proliferation Assessment | 4 weeks of treatment
  Analyzed in blood sampling.
Cytokine and Cortisol Assessment | 4 weeks of treatment
  Analyzed in blood sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Kleiner AFR, Souza Pagnussat A, Pinto C, Redivo Marchese R, Salazar AP, Galli M. Automated Mechanical Peripheral Stimulation Effects on Gait Variability in Individuals With Parkinson Disease and Freezing of Gait: A Double-Blind, Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Dec;99(12):2420-2429. doi: 10.1016/j.apmr.2018.05.009. Epub 2018 Jun 11. PMID 29902470